CLINICAL TRIAL: NCT01822457
Title: Effect of Nike FuelBand on Exercise and Function in Claudicants; a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12 LO 1896
Record Dates: First submitted 2013-02-19; First posted 2013-04-02 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Vascular Disease; Intermittent Claudication
Keywords: Peripheral vascular disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nike FuelBand (NFB) (Experimental): Patients will receive a Nike Fuel Band to encourage exercise.
  Interventions: Device: Nike FuelBand (NFB)
- control (No Intervention): Standard follow-up

INTERVENTIONS:
Device: Nike FuelBand (NFB) — The Nike Fuel Band (NFB) is a wrist-worn sensor with a built-in accelerometer for motion quantification. It is programmed to estimate the number of steps taken per day, and also predict energy expenditure in units known as Nike Fuel. Accompanying software allows the user to set daily targets and monitor their activity through a graphical user interface.
  Arms: Nike FuelBand (NFB)

SUMMARY:
This is a randomised controlled study of patients suffering from intermittent claudication (IC), to assess the impact of wearing a Nike FuelBand (NFB) on walking distances, exercise levels and quality of life.

DETAILED DESCRIPTION:
IC manifests as pain in the calf, thigh or buttock muscles when walking. It is caused by narrowing or blockage of the blood vessels in the legs.

The NFB is a discrete wristband with a built-in accelerometer to measure motion. It provides estimates of the number of steps taken and the amount of distance covered each day.

This study will be conducted over a period of 18 months at Imperial College Trust's vascular outpatients service. Patients that meet the inclusion/exclusion criteria will be asked to consider participating. Participants will receive routine diagnostic work up with the addition of having their walking distances measured on a lab treadmill. They will also have their functional status and mood assessed using a questionnaire. These assessments will be carried out a total of five times over the course of the study. Patients will not need to make any additional visits to hospital.

Patients will be randomly allocated to either the NFB group or the control group. Patients in the NFB group will be given a FuelBand with instructions on how to use it. All patients will be given routine instructions on maintaining activity and target daily walking distances. Target walking distances will be programmed into the NFB. Patients in the NFB group will be asked to record estimates of how far they have walked each day directly from their band. All patients will be contacted by telephone at a pre-arranged time to collect recordings.

Patients will be followed up at their routine 3-month follow up appointment and additionally at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80
* Referred to vascular rehabilitation service at St Marys Hospital (UK)
* IC involving the calf muscles
* Clinical and duplex investigations indicate Superficial Femoral Artery stenosis or occlusion

Exclusion Criteria:

* Clinical and duplex investigations indicate iliac disease
* Major joint disease in lower limb or lumbar spine/entrapment syndrome
* Significant cardiopulmonary limitations (NYHA>1)
* Maximum walking distance >500m
* Hospital inpatient/ living in a care home
* *Unfamiliarity with required technology
* History of dementia
* Unable to mobilize independently (does not include walking aids)
* IC not limiting factor of mobilization, limited by other medical problems
* Unable to attend supervised exercise programme
* Patient owns or uses any type of activity monitor
* Uses a walking frame *Patients should be able to use the NFB technology with minimal assistance

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Darzi, MD, FRCS, FRS, Principal Investigator — Imperial College NHS Healthcare Trust; Nicholas J Cheshire, MD, FRCS, Study Director — Imperial College NHS Healthcare Trust; Colin D Bicknell, MD, FRCS, Study Director — Imperial College NHS Healthcare Trust; Celia Riga, MD, FRCS, Study Director — Imperial College NHS Healthcare Trust
Locations (1):
- Imperial College NHS Healthcare Trust- St Marys, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nike FuelBand (NFB) | Control
Started | 20 | 17
Completed | 16 | 12
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nike FuelBand (NFB) | Control | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (10.3) | 70.7 (10.8) | 69.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 18 | 12 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Maximum Walking Distances
Description: Standardised treadmill test at the end of the study period
Time Frame: 12 months
Measure: Mean (Inter-Quartile Range); unit: Meters
Arm/Group | Nike FuelBand (NFB) | Control
Number analyzed (Participants) | 16 | 12
Meters | 147 [135 to 405] | 68 [40 to 75]

2. Secondary Outcome: Pain Free Treadmill Walking Distance
Description: Standardised treadmill test - first recognition of pain as reported by the patient.
Time Frame: 12 months
Measure: Mean (Inter-Quartile Range); unit: Meters
Arm/Group | Nike FuelBand (NFB) | Control
Number analyzed (Participants) | 16 | 12
Meters | 110 [55 to 200] | 44 [30 to 75]

3. Secondary Outcome: Disease Specific Quality of Life
Description: Assessed using VascuQol (Vascular Quality of life) Questionnaire score, range from 0 to 24, and higher value indicates a better health status.
  Each question has a four-point response scale (1 most problems - 4 no problems)
Time Frame: 12 months
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Nike FuelBand (NFB) | Control
Number analyzed (Participants) | 16 | 12
score on a scale | 5.8 [5.0 to 7.0] | 3.3 [2.4 to 4.6]

4. Secondary Outcome: Mood
Description: Assessed using the Hospital Anxiety and Depression Scale score, participants reply that is closest to how they have been feeling in the past months. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Score 0 to 3, 3 - Most of the time, 0 - Not at all.
Time Frame: 3 months
Population: Data not collected
Arm/Group | Nike FuelBand (NFB) | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Nike FuelBand (NFB) | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes